CLINICAL TRIAL: NCT03597217
Title: A Phase 1, 2-part Study Of Pf-05221304 In Healthy Japanese Adults: Part 1 - Randomized, Double-blind, Crossover, Single Dose Assessment Of Pharmacokinetics And Safety; Part 2- Randomized, Double-blind, Placebo-controlled, Multiple Dose Assessment Of Safety, Tolerability And Pharmacokinetics Of Pf-05221304
Brief Title: A Single and Multiple Dose Study of PF-05221304 in Healthy Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C1171013
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: PF-05221304, PK, Japanese, NASH, ACC inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A_Active (Experimental): 3 single doses treatment of PF-05221304
  Interventions: Drug: PF-05221304
- Cohort B_Active (Experimental): Repeated doses of PF-05221304
  Interventions: Drug: PF-05221304
- Cohort B_Placebo (Placebo Comparator): Repeated doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05221304 — 3, 10, 50 mg
  Arms: Cohort A_Active
Drug: PF-05221304 — 50 mg multiple dose
  Arms: Cohort B_Active
Drug: Placebo — Placebo
  Arms: Cohort B_Placebo

SUMMARY:
The current study is designed to evaluate the safety, tolerability and pharmacokinetics of PF-05221304 in healthy Japanese adult subjects following single and multiple dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects who, at the time of screening, are between the ages of 20 and 55 years, inclusive.
* Body mass index (BMI) of 17.5-30.5 kg/m2 inclusive; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) or clinical findings at Screening.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Cohort A: Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration (AUClast) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Maximum observed plasma concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Time to reach Cmax (Tmax) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Area under the plasma concentration time profile from time zero extrapolated to infinite time (as data permit) (AUCinf) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Terminal half life (as data permit) (t1/2) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Apparent clearance (as data permit) (CL/F) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort A: Apparent volume of distribution (as data permit) (Vz/F) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment of adverse events (AEs), clinical laboratory tests, vital signs (including blood pressure and pulse rate) and 12 lead ECG.

SECONDARY OUTCOMES:
Cohort A: Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment of adverse events (AEs), clinical laboratory tests, vital signs (including blood pressure and pulse rate) and 12 lead ECG.
Cohort B: Area under the plasma concentration time profile from time zero to time τ (tau), the dosing interval (ACUtau)(Day 1) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 hours post dose
Cohort B: Area under the plasma concentration time profile from time zero to time τ (tau), the dosing interval (ACUtau)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Maximum plasma concentration during the dosing interval (Cmax)(Day 1) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 hours post dose
Cohort B: Maximum plasma concentration during the dosing interval (Cmax)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Time to reach Cmax (Tmax)(Day 1) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 hours post dose
Cohort B: Time to reach Cmax (Tmax)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Minimum plasma concentration during the dosing interval (Cmin)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Peak trough ratio (PTR)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Observed accumulation ratio (Rac)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Observed accumulation ratio for Cmax (Rac,Cmax)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Terminal half life (t1/2)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Apparent volume of distribution (Vz/F)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose
Cohort B: Apparent clearance (CL/F)(Day 14) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Keikokai Medical Corporation, Hachioji-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171013&StudyName=A+Phase+1%2C+2-part+Study+Of+Pf-05221304+In+Healthy+Japanese+Adults%3A+Part+1+-+Randomized%2C+Double-blind%2C+Crossover%2C+Single+Dose+Assessment+Of+Pharmacokinetics+And+Safety%3B+Part+2-+Randomized%2C+Double-blind%2C+Placebo-controlled%2C+Multiple+Dose+Assessment+Of+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Pf-05221034
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171013&StudyName=A+Phase+1%2C+2-part+Study+Of+Pf-05221304+In+Healthy+Japanese+Adults%3A+Part+1+-+Randomized%2C+Double-blind%2C+Crossover%2C+Single+Dose+Assessment+Of+Pharmacokinetics+And+Safety%3B+Part+2-+Randomized%2C+Double-blind%2C+Placebo-controlled%2C+Multiple+Dose+Assessment+Of+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Pf-05221304